

NCT03310723

10/23/2019

Study was approved by the University of British Columbia Children's and Women's Research Ethics Board

Inclusion criteria: healthy, term (≥ 36 weeks gestation), non-labouring parturients admitted for elective caesarean delivery or induction of labour

Exclusion criteria: ASA physical status 3 or above; any medical condition that could affect gas exchange; BMI ≥ 40 kg/m²; known airway pathology; obstructed nasal airway; or unable to tolerate a tight-fitting facemask.

Microsoft Excel 2010 was used to generate a randomisation sequence with 1:1 allocation to either HFNO or control groups.

All patients were first placed in a 30-degree head up position using the Troop<sup>™</sup> (Goal Medical, LLC, Eugene, OR, USA) elevation pillow and with a right lateral pelvic wedge to minimise aortocaval compression. A nose clip was applied and each patient was asked to breathe 21% oxygen at 12 l.min<sup>-1</sup> through a standardised mouthpiece using tidal volume breathing. The mouthpiece was connected to an anaesthetic circle system with a two-litre reservoir bag, heat moisture exchange filter and an oxygen analyser. At the end of 30 s, baseline values for oxygen saturation, respiratory rate, heart rate and EtO₂ were recorded.

Patients in the standard oxygen flow rate facemask group (control) were then pre-oxygenated with 100% oxygen, using tidal volume breathing and a tight-fitting facemask attached to a circle system, with an oxygen flow rate of 15 l.min<sup>-1</sup>. End-tidal carbon dioxide waveform analysis was monitored to ensure a tight seal was achieved between the patient and the facemask. After 3 min, patients were asked to hold their breath for a few seconds and the nose clip was re-attached. The patients then exhaled fully and continued to breathe for several breaths via the mouthpiece (delivering 21% oxygen) to ensure the highest value for EtO<sub>2</sub> was measured.

Patients in the HFNO group were pre-oxygenated with 100% oxygen using tidal volume breathing and the Optiflow™ HFNO nasal high-flow cannula system (Fisher and Paykel Healthcare Ltd, Auckland, New Zealand). The oxygen flow rate was initially started at 30 l.min⁻¹and gradually increased to a maximum of 70 l.min⁻¹ over the first 30 s. If a patient did not tolerate the flow rate, it was

reduced to a level the patient could tolerate, typically 50–60 l.min<sup>-1</sup>. Patients were specifically instructed to breathe via their nose with a closed mouth and the percentage of time this was achieved was recorded (0%, 25%, 50% or 100%). After 3 min, the patients were asked to hold their breath for a few seconds while the HFNO was quickly removed and the nose clip re-attached. The patients then exhaled fully and continued to breathe for several breaths via the mouthpiece (delivering 21% oxygen) to ensure the highest value for EtO<sub>2</sub> was measured.

Patients in both groups then underwent a washout period for up to 5 min until the EtO<sub>2</sub>returned to within 10% of their baseline value. Once washout was completed, both groups repeated 30 s of tidal volume breathing followed by eight vital capacity breaths using their respective pre-oxygenation methods. During the initial 30 s of tidal volume breathing, the oxygen flow rate in the HFNO group was increased from 30 to 70 l.min<sup>-1</sup> and EtO<sub>2</sub> was measured at the conclusion of eight vital capacity breaths. The time taken to complete 30 s of tidal volume breathing and eight vital capacity breaths was also recorded.

Immediately after the study, patient satisfaction was assessed using a 5-category Likert scale for acceptability (acceptable, slightly acceptable, neutral, slightly unacceptable or unacceptable) and comfort (completely comfortable, slightly comfortable, neutral, slightly uncomfortable or completely uncomfortable).

## **Outcomes**

The primary outcome was EtO<sub>2</sub> after pre-oxygenation, with factorial comparisons also being made between HFNO and standard flow rate facemask, and also between 3 min of tidal volume breathing and eight vital capacity breaths.

The Secondary outcomes were the proportion of patients achieving an  $EtO_2 \ge 90\%$ , percentage of time patients had their mouths closed during HFNO pre-oxygenation and tolerability (comfort and acceptability) of both pre-oxygenation techniques.

## Sample Size Calculation

The study sample size was determined based on a prior study demonstrating that the mean (SD) EtO<sub>2</sub> achieved following 3 min of pre-oxygenation in healthy, non-pregnant subjects with HFNO and facemask was 85.6% (6.4%) and 88.5% (6.2%), respectively. We initially powered the study for a non-inferiority comparison. The criterion for non-inferiority with respect to EtO<sub>2</sub> concentration achieved after 3 min was considered to have been met if the upper limit of a two-sided 95%CI for the absolute difference of EtO<sub>2</sub> concentration between groups was less than 10%. Using a non-inferiority design, assuming a non-inferiority margin of 10 and a standard deviation of 6.3, and that the HFNO group would have a mean approximately 3% lower than the control group, 26 patients (13 per group) were required to achieve a power of 90% with a type-1 error of 0.05. To account for attrition and study dropouts due to equipment errors (i.e. lack of a tight seal for waveform analysis), the sample size was increased to 40 (20 per group).

After patient recruitment we realised that as a physiological and not clinical study. a standard superiority design was more appropriate. Using a superiority analysis with 20 patients per group there would have been approximately 31% power to detect a difference in means of 3% with a standard deviation of 6.3. Consequently, data for primary outcomes were analysed using mixed-effects linear regression. Mixed-effects models take into account the repeated-measures aspect of the data and control for correlations among measurements from the same patient. To determine if there was a difference in how the treatment groups responded, we tested for an interaction term between group and time-point. If a significant interaction was found, we followed it up with pairwise tests of the estimated marginal means between the groups at each time-point (e.g. HFNO baseline vs. control baseline) using the Kenward-Roger method to estimate confidence intervals, and controlling for multiple comparisons using Tukey's method. The proportion of patients achieving an EtO<sub>2</sub>  $\geq$  90%, comfort and acceptability was compared using Fisher's exact test. A p value < 0.05 was considered statistically significant. Statistical analysis was performed using RStudio version 1.0.153 (Integrated Development for R. RStudio, Inc., USA; http://www.rstudio.com) and R version 3.4.1, release date June 30, 2017 (The R Foundation for Statistical Computing, Austria).